CLINICAL TRIAL: NCT00958867
Title: Enhancing Cognition and Functional Independence in Senior Women With Mild Cognitive Impairment: A Randomized Trial of Aerobic vs. Resistance Training
Brief Title: EXCEL: Exercise for Cognition and Everyday Living for Seniors With Memory Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Pacific Alzheimer Research Foundation (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H09-00365
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Resistance exercise training; aerobic exercise training
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Six-month, twice-weekly aerobic training (AT) program
  Interventions: Behavioral: Exercise program (AT)
- 2 (Experimental): Six-month, twice-weekly resistance training (RT) program
  Interventions: Behavioral: Exercise training (RT)
- 3 (Active Comparator): Six-month, twice-weekly stretch & relax (S & R; control) program
  Interventions: Behavioral: Exercise training (S & R; control)

INTERVENTIONS:
Behavioral: Exercise program (AT) — Six-month, twice-weekly aerobic training (AT) program
  Arms: 1
Behavioral: Exercise training (RT) — Six-month, twice-weekly resistance training (RT) program
  Arms: 2
Behavioral: Exercise training (S & R; control) — Six-month, twice-weekly stretch & relax (S & R; control) program
  Arms: 3

SUMMARY:
Alzheimer's disease (AD) is a major health issue in Canada; it affects over 8% of the population aged over 65 years. Persons with AD have a reduced quality of life as they become dependent on others for activities of daily living (ADLs). This problem of loss of independence - functional dependence - is one focus of this grant application. It is projected that by 2020, Canada will have well over 10 million seniors with moderate to severe functional dependence. Functional dependence was the most significant contributor to an annual cost of dementia that had already reached $4 billion in the 1990s.

Mild cognitive impairment (MCI) is a well-recognized risk factor for both AD and functional dependence. Within the broader assessment of cognitive function, the literature suggests that executive functioning - the ability to concentrate, to attend selectively, to plan and strategize - is a robust cognitive predictor of functional status in seniors. Specifically, Royall and colleagues demonstrated executive functioning independently explained 43% of the functional status in community-dwelling seniors dementia. The researchers will investigate executive functioning in seniors with MCI.

Randomized trials of various exercise interventions have proven that exercise has many systemic benefits. Data are emerging that physical activity may improve cognition - specifically executive function - in healthy adults. The researchers' own pilot data suggest that resistance training in seniors may improve executive functioning as assessed by neuropsychological tests and neuro-imaging. However, at present the Cochrane Database of Systematic Reviews indicates there are insufficient published data to guide exercise prescription to prevent AD. In persons with MCI, no published studies have reported on whether physical activity can improve executive function, or delay its decline and thus, prevent or delay the onset of functional dependence (and later, dementia).

Therefore, among seniors with MCI, the researchers will investigate whether or not specific exercise prescription can: 1) provide absolute or relative improvement in cognitive function, particularly executive function; and 2) help maintain functional independence. This will facilitate the development of effective exercise-based strategies for the prevention of both cognitive and functional decline in the large population of seniors with MCI - people at greatly increased risk for AD.

The researchers' proposed research aims to ascertain whether a six-month, twice-weekly aerobic training (AT) program and a six-month, twice-weekly resistance training (RT) program, compared with a six-month, twice-weekly stretch & relax (S & R; control) program, will significantly improve cognition and functional status in community-dwelling women with MCI aged 70 years and older.

Primary Hypothesis:

At the end of six-month randomized trial, compared with the S & R program, both the AT and RT programs will significantly improve cognitive performance, as assessed by neuropsychological testing.

Secondary Hypotheses:

At the end of the six-month randomized trial, compared with the S & R program, participants of the AT and RT programs will:

1. Demonstrate evidence of cortical plasticity by fMRI, such as increased activation in cortical regions responsible for item and relational memory; and
2. Will significantly improve their everyday problem solving ability.

DETAILED DESCRIPTION:
STUDY DESIGN, TRIAL PROFILE, AND TIMELINE To achieve our research objectives, we will conduct a six-month, single-blinded (assessors), randomized trial. 75 community-dwelling older women with MCI will be randomly assigned to one of three experimental groups: 1) RT; 2) AT; or 3) S & R (Control). The study sample is restricted to women as the magnitude of response in cognition to exercise differs between sexes.

METHODS Recruitment We will recruit seniors who are interested in a study of exercise and cognition through media such as newspaper ads, flyers, and posters in community and senior centres. Interested individuals be screened. The screening session will include the following: 1) MMSE ; 2) Montreal Cognitive Assessment (MoCA) ; and 4) Lawton and Brody Instrumental Activities of Daily Living Scale. Individual who meet the inclusion criteria will be invited to join the research study.

Inclusion Criteria

1. Community-dwelling senior women as the female to male ratio for dementia is 2:1;
2. Aged 70 years and older;
3. Subjective memory complaints as determined by interview;
4. MMSE score > 24;
5. Scored < 26 on the MoCA;
6. Visual acuity of at least 20/40, with or without corrective lenses; and
7. Physician approval for participation in an exercise program. Exclusion Criteria

1) Diagnosed neurodegenerative disease (e.g., AD) and stroke; 2) Have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease; 3) Diagnosed with a psychiatric condition; 4) Previously diagnosed with dementia of any type; Measurements We have extensive experience in using each of the following methods and instruments. All measures, unless otherwise indicated, will be assessed at each measurement session.

General Screen and Descriptors (90 mins)

1. General Health and Socioeconomic Status: General health and socioeconomic status will be ascertained by a questionnaire.
2. Global Cognitive Function and Depression: Global cognitive function will be assessed using the MMSE. The Beck's Depression Inventory (BDI) will be administered. MCI Screen: There are no consensus criteria for the clinical classification of MCI. The MoCA will be used to screen participants for MCI. The MoCA is a brief screening tool for MCI with high sensitivity and specificity. It is a 30-point test covering eight cognitive domains and scores below 26 are considered to be abnormal. A bonus point is given to those with less than 12 years of education.
3. Physical Activity Level: Physical activity, not including the study-assigned exercise classes, will be determined at baseline and throughout the six-month study period. We will administer the valid and reliable Physical Activities Scale for the Elderly (PASE) questionnaire monthly. Designed for those aged 65 years and older, participants use a 12-item scale to self-report the average number of hours per day spent participating in leisure, household, and occupational physical activities over the previous seven-day period.
4. IADLs: Participants will complete the Lawton and Brody Instrumental Activities of Daily Living Scale to screen for impaired IADLs. This scale subjectively assesses ability to telephone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibility for own medication, and ability to handle finances.

Cognitive Performance Measures:

Memory:

We will assess item and relational memory using a computerized paradigm. We will also assess spatial memory and working memory (i.e., N-1 back) using computer paradigms. In all computer paradigms, we will record reaction time and accuracy. We will use the RAVLT to assess verbal memory.

Executive Functions:

We will assess three executive functions: 1) set shifting using the Trail Making Test (Part B) and a computerized paradigm of dual-task; 2) updating (i.e., working memory) using the verbal digits backward test and a computerized paradigm of N-back; and 3) response inhibition using the Stroop Colour-Word Test.

Cortical Activation (60 mins): To accurately assess the effect of both AT and RT on cortical plasticity, we will collect pre- and post-intervention fMRI data from all participants (i.e., AT, RT, and S & R).

Muscular Strength: We will assess dominant quadriceps (isometric) strength by strain gauge to the nearest 0.5 kilogram.

Six-Minute Walk (6 MWT): This is a walking test of physical status to assess general cardiovascular capacity in seniors 19. The total distance walked in meters in six minutes is recorded.

Balance and Mobility: General balance and mobility will be assessed with the National Institute on Aging (NIA) Balance Scale.

Everyday Problem Solving Ability will be assessed using Everyday Problems Test (EPT). The EPT is a research and assessment tool for measuring adults' ability to solve tasks of daily living that involve printed material. The focus of the measure is on assessing the adults' cognitive competence to reason and solve problems associated with daily living.

Randomization After baseline measurement, participants will be randomized by computer generated random draw to one of the three experimental groups (AT, RT, and S & R) using www.randomization.com.

Exercise Programs Resistance Training: The protocol for the RT program will be progressive and high-intensity with the aim of increasing muscle strength in the extremities and the trunk. Both a Keiser® Pressurized Air system (Keiser Corp.CA, US) and free weights will be used to provide the training stimulus. Participants will undergo a two-week familiarisation period with the equipment and the exercises. The exercises will consist of biceps curls, triceps extension, seated row, latissimus dorsi pull downs, mini-squats, mini-lunges, hamstring curls, and calf raises. The intensity of the training stimulus will initially be at 50% to 60% of 1 repetition maximum (RM) as determined at week two, with a work range of two sets of 10-15 repetitions and progress to 75% to 85% of 1RM at a work range of six to eight repetitions (two sets) by week four. The training stimulus will be increased using the 7RM method, when two sets of 6-8 repetitions are completed with proper form and without discomfort. Squats and lunges will be performed initially with body weight; loading will be increased only when proper form is maintained for two sets of 10 repetitions. The number of sets completed and the load lifted for each exercise will be recorded for each participant at every class.

Cardiovascular Training: The AT program will be an outdoor walking program. We will use three techniques to monitor exercise intensity. Each participant will: 1) wear a heart rate monitor and will be asked to work at 65% to 80% of her age specific target heart rate; 2) subjectively monitor the intensity of each workout using the Rating of Perceived Exertion.

Stretch and Relax (Control): The S &R program will consist of stretching exercises, deep breathing, and relaxation techniques. There is no evidence that these exercises improve cognitive function. This group will serve to control for confounding variables such as physical training received by traveling to the community centre for twice-weekly classes, social interaction, and changes in lifestyle secondary to study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling senior women;
2. Aged 70 years and older;
3. Subjective memory complaints as determined by interview;
4. MMSE score > 24/30;
5. Scored < 26/30 on the MoCA (74);
6. Visual acuity of at least 20/40, with or without corrective lenses; and
7. Physician approval for participation in an exercise program.

Exclusion Criteria:

1. Diagnosed neurodegenerative disease (e.g., AD) and a history of stroke;
2. Have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease;
3. Diagnosed with a psychiatric condition; or
4. Diagnosed with dementia of any type.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Cognitive performance after 3 and 6 months of training | 6 months

SECONDARY OUTCOMES:
Everyday problem-solving ability after 3 and 6 months of exercise training, brain function after 6 months of training and physical function after 3 and 6 months of training | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, PT, Principal Investigator — teresa.ambrose@ubc.ca
Locations (1):
- Centre for Hip Health Mobility, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] ten Brinke LF, Bolandzadeh N, Nagamatsu LS, Hsu CL, Davis JC, Miran-Khan K, Liu-Ambrose T. Aerobic exercise increases hippocampal volume in older women with probable mild cognitive impairment: a 6-month randomised controlled trial. Br J Sports Med. 2015 Feb;49(4):248-54. doi: 10.1136/bjsports-2013-093184. Epub 2014 Apr 7. PMID 24711660
- [Derived] Davis JC, Bryan S, Marra CA, Sharma D, Chan A, Beattie BL, Graf P, Liu-Ambrose T. An economic evaluation of resistance training and aerobic training versus balance and toning exercises in older adults with mild cognitive impairment. PLoS One. 2013 May 14;8(5):e63031. doi: 10.1371/journal.pone.0063031. Print 2013. PMID 23690976